CLINICAL TRIAL: NCT02376738
Title: Regional Activation of Leukocytes in Coronary Artery Disease
Acronym: REAL-CAD
Status: Completed | Type: Observational
Sponsor: Sint Franciscus Gasthuis (Other)
Responsible Party: Principal Investigator, M.A. de Vries, PhD Student, Sint Franciscus Gasthuis
Other Study IDs: REAL-CAD
Record Dates: First submitted 2015-02-18; First posted 2015-03-03 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-02

CONDITIONS: Inflammation; Coronary Artery Disease
MeSH Terms: conditions — Inflammation; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to evaluate the role of leukocyte activation in coronary artery disease

DETAILED DESCRIPTION:
1. The primary aim of REAL CAD is to determine regional differences of leukocyte activation in different vascular beds in vivo.
2. The secondary aim is to investigate differences in leukocyte activation between diabetic and CAD subjects and patients suffering from both.
3. The third aim is to investigate the relationship between complement components, triglycerides and leukocyte activation markers in order to gain more insight into the causative processes leading to activation of leukocytes.
4. The fourth aim is to get more insight in the MBL genotypes and serum levels of CAD and/or diabetic patients and the 'healthy' groups included in our study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects scheduled to undergo a coronary catheterization
* Provide written informed consent
* Aged >18 and <75 years
* BMI < 35 kg/m2

Exclusion Criteria:

* Emotionally and intellectually not capable to decide about participation in the study and the consequences of participation. Subjects who are not able to understand the patient information
* CRP > 20 mg/l
* Unstable angina pectoris
* CABG or PTCA during the last 6 months
* Alcohol use > 2 units/day
* Aberrations in kidney, liver and thyroid function
* Use of any experimental medication within 6 months of the catheterization
* The use of immunosuppressive drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing coronary angiography
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2007-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Assess the level of leukocyte activation in different vascular beds, by measuring monocyte CD11b and neutrophil CD11b and CD66b in blood obtained from the left and right coronary artery, the abdominal aorta, the femoral artery and a peripheral vein | Baseline

SECONDARY OUTCOMES:
Investigate differences in leukocyte activation between patients with and without diabetes mellitus or coronary artery disease by comparing the level of monocyte CD11b and neutrophil CD11b and CD66b | Baseline
To investigate the predictive value of leukocyte activation markers CD11b and CD66b in different vascular regions in the prediction of future coronary events, by measuring these markers at baseline | 6 years follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Castro Cabezas, MD PhD, Principal Investigator — Sint Franciscus Gasthuis
Locations (1):
- Sint Franciscus Gasthuis, Rotterdam, South Holland, Netherlands